CLINICAL TRIAL: NCT03493724
Title: Interest of the Photographs by Smartphone During the Requests of Opinion Specialized in the Department of Dermatology of the CHRU of Nancy
Brief Title: Interest of Photographs by Smartphone in Dermatology
Acronym: PHOTODERM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-A02607-46
Record Dates: First submitted 2018-03-09; First posted 2018-04-10 (Actual); Last update posted 2018-04-10 (Actual); Status verified 2018-02

CONDITIONS: Dermatitis
MeSH Terms: conditions — Dermatitis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No

INTERVENTIONS:
Other: telemedecine — to evaluate the diagnostic performance of the photographs made by Smartphone, during requests for emergency dermatological advice
  Other Names: evaluation of photographs in dermatology

SUMMARY:
To study the diagnostic performance of the images on the smartphone compare the result of the clinical examination, all the dermatoses combined and by family of pathology (inflammatory, wound, oncology, infectious, allergology), during urgent request requests in dermatology

DETAILED DESCRIPTION:
The study is conducted in the dermatology department, for a maximum duration of 6 months. We include patients who require dermatological advice and for whom their doctor sends us photographs.

Doctors contact us by telephone, describe the symptoms and send photographs according to the secure procedure.

Patients are admitted for consultation and the diagnosis by photography is compared with the clinical diagnosis

ELIGIBILITY:
Inclusion Criteria:

* For which our fellow doctors ask a dermatological opinion for diagnostic purposes, after clinical examination of the patient, in an emergency
* After obtaining the oral consent by the requesting doctor then informing and signing a non-opposition form during the consultation at the University Hospital of Nancy
* Affiliation to a social protection
* Doctors must have signed and sent back an ethical charter, where they undertake to send the image via MSsante, then to erase the image of the smartphone

Exclusion Criteria:

* Patients under the protection of justice, tutorship or curatorship
* Doctors : lack of smartphone powerful enough to offer a quality image

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Major patients presenting with dermatitis, requiring specialized advice in dermatology at the University Hospital of Nancy
Sampling Method: Probability Sample
Enrollment: 205 (Estimated)
Dates: Start 2018-02-13 (Actual); Primary Completion 2018-07-01 (Estimated); Study Completion 2018-09-01 (Estimated)

PRIMARY OUTCOMES:
sensitivity, specificity, positive and negative predictive values globally | through study completion, an average 6 months
  evaluation of the diagnostic performance of the test
sensitivity, specificity, positive and negative predictive values stratified | through study completion, an average 6 months
  stratified on the families of pathologies : infectious pathology, inflammatory dermatosis, allergology, wound, oncology

SECONDARY OUTCOMES:
Calculation of Cohen's kappa concordance between dermatologists | through study completion, an average 6 months
  assessment of interobserver diagnostic agreement

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU Nancy, hopitaux de Brabois, Nancy, Vandoeuvre Les Nancy, France

IPD SHARING:
Plan to Share IPD: No